CLINICAL TRIAL: NCT07309224
Title: Employing Peer Outreach and Whole Health in Recovery (EMPOWER) for Homeless-Experienced Veterans: A Hybrid Type III Implementation Trial (QUE 25-014)
Brief Title: Employing Peer Outreach and Whole Health in Recovery for Homeless-Experienced Veterans
Acronym: EMPOWER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 26-002
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorder; Mental Health Disorder; Homelessness
Keywords: Veterans; Homeless Persons; Peer Influence; Whole Person Health; Implementation Science
MeSH Terms: conditions — Substance-Related Disorders; Mental Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Intervention Model Description: The investigators will conduct an adaptation of the multi-site hybrid III cluster randomized trial design to evaluate the implementation of EMPOWER through tailored low-intensity and high-intensity strategies. Specifically, the investigators will use a staircase design - an adaptation to stepped wedge designs (SWD). This design accommodates more flexible implementation (i.e., less burden to sites and clinicians) while at the same time offering robust statistical efficiency, given that statistical information is often strongest around time periods in the SWD when a strategy switches. For EMPOWER, of interest is the effect of switching from Low Intensity (LI - i.e., Audit and Feedback) to High Intensity (HI - i.e., Facilitation) implementation strategies; an imbalanced design will be employed in which sites will spend twice as long in HI than LI (12 months vs. 6 months, respectively).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-Intensity (LI) (Active Comparator): For the LI phase of a site's implementation, a light-touch strategy will be used to implement EMPOWER; specifically, Audit and Feedback. In Audit and Feedback, key stakeholders at sites receive summarized data about their performance relative to a standard or benchmark. Specifically, HUD-VASH peers and supervisors at each site will be emailed monthly automated reports on EMPOWER fidelity data from the EHR (e.g., % of HUD-VASH patients with a Personal Health Plan note) as well as aggregated data on treatment engagement via the Hot Spot dashboard (e.g., % of HUD-VASH Veterans with an SUD diagnosis who received SUD specialty care in the past month). The monthly reports will include tailored action item recommendations based on the local site's performance. Under the LI strategy, sites will not be provided interactive support to review these reports.
  Interventions: Behavioral: Employing Peer Outreach and Whole Health in Recovery (EMPOWER)
- High-Intensity (HI) (Experimental): For the HI phase of a site's implementation, a higher-intensity strategy will be used to implement EMPOWER; specifically, Facilitation. Facilitation is a collaborative strategy in which trained individuals work with organizations or teams to support the adoption, implementation, and sustainment of an evidence-based practice (EBP). It is a dynamic process that involves tailored guidance, problem-solving, technical assistance, and capacity-building activities to address specific barriers and leverage facilitators of change. To this end, external facilitators often collaborate with local champions to bring expertise regarding the implementation processes and have transferable knowledge in relevant clinical and behavior change models that inform the EBP's implementation.
  Interventions: Behavioral: Employing Peer Outreach and Whole Health in Recovery (EMPOWER)

INTERVENTIONS:
Behavioral: Employing Peer Outreach and Whole Health in Recovery (EMPOWER) — EMPOWER is a multicomponent intervention to facilitate homeless-experienced veterans' (HEVs) care engagement: (DATA ANALYTICS) HUD-VASH case managers identify high-need, HUD-VASH Veterans on the Homeless Registry Hot Spot Report. Veterans' profiles are reviewed to learn about their chronic health conditions, housing status, acute care use, and engagement in supportive care. (PEER SUPPORT): HUD-VASH peers meet with identified Veterans for up to six months, averaging once-per week sessions for the first three months, with step-down in frequency as Veterans begin to engage in services and reach their goals. (WHOLE HEALTH): During sessions, peers use a Whole Health approach to collaboratively develop personal health goals that align with the Veteran's priorities and values-e.g, help Veterans completing a Personal Health Inventory and developing a Personal Health Plans. Provider communications: Peers communicate with a Veteran's care providers to share the Veteran's personal health goals.
  Other Names: EMPOWER

SUMMARY:
Homelessness is a national crisis in the United States, particularly in the veteran population. Due to multiple chronic conditions, homeless individuals frequently become hospitalized or are treated in emergency departments. Care engagement can mitigate this risk. Interventions grounded in evidence-based practices of peer support and whole health are effective for increasing care engagement. However, implementation of such interventions with high-acuity patients often requires strategies that are intensive and costly. This trial will evaluate the relative impacts and costs of using a high-intensity (vs. low-intensity) strategy to implement a peer-led, whole health intervention for homeless-experienced veterans in permanent supportive housing.

DETAILED DESCRIPTION:
Background: Homelessness is a national crisis in the United States, particularly in the Veteran population. Due to multiple chronic conditions, homeless individuals have elevated risk for acute care service use. Engagement in primary and specialty care can mitigate this risk. Interventions grounded in evidence-based practices of peer support, patient-centered care, and whole health are effective for increasing service engagement. However, implementation of such interventions with high-acuity patients often requires multi-component strategies that are intensive and costly. This study protocol describes a hybrid type 3 effectiveness-implementation trial of Employing Peer Outreach and Whole Health in Recovery (EMPOWER) with high-need, homeless-experienced Veterans in permanent supportive housing and will evaluate the impact and cost of a high-intensity (vs. low-intensity) strategy on implementation outcomes.

Methods: (Aim 1) At 7 sites in the Veterans Health Administration (VA), a mixed methods pre-implementation evaluation will identify determinants and their potential impact on uptake of the EMPOWER and inform modifications to the intervention and implementation strategies as needed. (Aim 2) A staircase cluster randomized design will evaluate the rollout of the implementation strategies, beginning with Audit and Feedback (low-intensity) and then switching to Facilitation (high-intensity) after 6 months. Facilitation is hypothesized to have a greater impact on the reach, effectiveness, adoption, implementation (fidelity), and maintenance of EMPOWER. (Aim 3) A budget impact analysis will estimate the average cost of implementing EMPOWER at future sites and comparative costs for implementing the low- and high-intensity strategies.

Anticipated Impact: This study will provide information on the relative impacts and relative costs of strategies aimed at implementing a peer-led, patient-centered, whole health intervention for homeless-experienced Veterans in permanent supportive housing. The findings will provide guidance to VA and other healthcare systems that serve the aging population of homeless-experienced Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be identified from VA's Homeless Registry "Hot Spot" reports, which use real-time data on acute care service utilization to identify high-need, housing-insecure patients.
* These reports identify Veterans on the VA Homeless Registry (i.e., those who had received VA housing services in the past two years) who had >1 hospital admissions and/or >2 ED visits in the past quarter of the fiscal year.
* From these reports, the investigators will identify patients at each implementation site who are

  * (a) currently enrolled in HUD-VASH
  * (b) have a mental health and/or SUD diagnosis

Exclusion Criteria:

* Not flagged on the VA's Homeless Registry Hot Spot Report
* Not currently enrolled in HUD-VASH
* Does not have a mental health and/or substance use disorder diagnosis
* Is not a patient at a participating site of the implementation trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Reach | 18 months
  Reach will be measured in terms of the number of patients who are willing to receive EMPOWER, out of all patients that are estimated to be eligible at potential sites.
Adoption | 18 months
  Adoption will be measured in terms of the number of peers in HUD-VASH at sites that are trained in EMPOWER and initiate the intervention with eligible patients at their site.
Implementation | 18 months
  Implementation will be measured in terms of rate of completion of peer encounters at the site level and rate of completion of the elements of EMPOWER (e.g., percentage of EMPOWER patients with a Personal Health Plan entered into the EHR; percentage of EMPOWER patients who were referred to a Whole Health service at the local facility). These rates will be measured via activity logs embedded in the EHR and electronic data capture logs to document type and length of encounters.
Maintenance | 18 months
  Maintenance will be measured by the number of patients who are continuing to engage in EMPOWER and other VA services over the duration of the implementation phase (18 months).

SECONDARY OUTCOMES:
Effectiveness - Mental Health Outpatient Care | 6 months
  Among patients who receive EMPOWER and have a mental health diagnosis, the number of outpatient visits for mental health care they receive after 6 months, as measured by VA administrative data (e.g., stop codes of outpatient encounters).
Effectiveness - Substance Use Disorder Outpatient Care | 6 months
  Among patients who receive EMPOWER and have a diagnosis of a substance use disorder (SUD), the number of outpatient visits for SUD care they receive after 6 months, as measured by VA administrative data (e.g., stop codes of outpatient encounters).
Effectiveness - Primary Care | 6 months
  Among patients who receive EMPOWER, the number of primary care visits they attend after 6 months, as measured by VA administrative data (e.g., stop codes of outpatient encounters).
Effectiveness - Whole Health care | 6 months
  Among patients who receive EMPOWER, the number of outpatient visits for Whole Health-related care they receive after 6 months, as measured by VA administrative data (e.g., stop codes of outpatient encounters of health coaching and other complementary and integrative services).
Effectiveness - Hospitalizations | 6 months
  Among patients who receive EMPOWER, the number of bed days of care for ambulatory-care sensitive conditions after 6 months, as measured by VA administrative data (e.g., Bedsection codes).
Effectiveness - ED visits | 6 months
  Among patients who receive EMPOWER, the number of visits to an emergency department after 6 months, as measured by VA administrative data (e.g., stop codes).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Blonigen, PhD MA, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No